CLINICAL TRIAL: NCT00849251
Title: Combination Pegylated Liposomal Doxorubicin, Bortezomib, Cyclophosphamide, and Dexamethasone for Multiple Myeloma (PLD-BCD)
Brief Title: Pegylated Liposomal Doxorubicin Hydrochloride, Bortezomib, Cyclophosphamide, and Dexamethasone in Treating Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: One of the study drugs is not available.
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pamela S Becker, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6817; NCI-2009-01665 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; liposomal doxorubicin; Bortezomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy and enzyme inhibitor) (Experimental): Patients receive cyclophosphamide IV or PO over 1 hour, bortezomib IV over 3 minutes, and dexamethasone IV or PO on days 1, 8, and 15. Patients also receive pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 8. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: bortezomib; Drug: dexamethasone

INTERVENTIONS:
Drug: cyclophosphamide — Given IV or PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: pegylated liposomal doxorubicin hydrochloride — Given IV
  Other Names: CAELYX; Dox-SL; DOXIL; doxorubicin hydrochloride liposome; LipoDox
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: dexamethasone — Given IV or PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pegylated liposomal doxorubicin hydrochloride and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Giving pegylated liposomal doxorubicin hydrochloride together with bortezomib, cyclophosphamide, and dexamethasone may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects of giving pegylated liposomal doxorubicin hydrochloride together with bortezomib, cyclophosphamide, and dexamethasone and to see how well it works in treating patients with multiple myeloma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine efficacy of this novel combination in newly diagnosed patients with multiple myeloma.

SECONDARY OBJECTIVES:

I. To determine the toxicity of this novel combination regimen in previously treated patients and newly diagnosed patients with multiple myeloma.

OUTLINE:

Patients receive cyclophosphamide intravenously (IV) or orally (PO) over 1 hour, bortezomib IV over 3 minutes, and dexamethasone IV or PO on days 1, 8, and 15. Patients also receive pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 8. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of treatment, patients are followed up every 3 months for 2 years, then annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Relapsed, refractory patients with multiple myeloma who have failed at least one prior regimen not including dexamethasone alone
* Cohort 2: Newly diagnosed patients with previously untreated multiple myeloma; prior dexamethasone permitted; not to exceed 320 mg
* Diagnosis of multiple myeloma with quantifiable monoclonal protein or light chain identified by serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP), or serum free light chain assay
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count >= 1.5
* Platelet count >= 75,000 unless slightly lower due to disease with the approval of the principal investigator (PI)
* Serum creatinine =< 2.0 mg/dL
* Serum bilirubin =< 1.2
* Aspartate transaminase (AST)/alanine transaminase (ALT) =< 2.5 x upper limit of normal (ULN)
* Alkaline phosphatase =< 2.5 x ULN
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Left ventricular ejection fraction greater than or equal to 50% by multi gated acquisition scan (MUGA)
* Female subjects must be post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study; female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Male patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol
* Use of other anticancer therapy within 15 days or before study entry; the patient must have recovered from all acute non-hematological toxicities from any previous therapy
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment, despite appropriate antibiotics or other treatment; for cardiac dysfunction, myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection) on antiviral, antibiotic and antifungal treatment
* Patient has >= Grade 2 peripheral neuropathy within 14 days before enrollment
* Patient has hypersensitivity to bortezomib, boron or mannitol
* Pregnant or lactating patients
* Cumulative dose of doxorubicin of 400 mg/m^2 or greater, or if this level would be exceeded during the current study
* Any significant concurrent illness, condition, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Have had a diagnosis of another malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy including the following:
* Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed;
* Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed;
* Prior autologous stem cell transplant (Cohort 2 only);
* Prior allogeneic stem cell transplant;
* Patient has received other investigational drugs within 14 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Becker, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Relapsed Disease (Cohort I): Patients with relapsed multiple myeloma receive cyclophosphamide IV or PO over 1 hour, bortezomib IV over 3 minutes, and dexamethasone IV or PO on days 1, 8, and 15. Patients also receive pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 8. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  cyclophosphamide: Given IV or PO
  pegylated liposomal doxorubicin hydrochloride: Given IV
  bortezomib: Given IV
  dexamethasone: Given IV or PO
- Newly Diagnosed Disease (Cohort II): Patients with newly diagnosed multiple myeloma receive cyclophosphamide IV or PO over 1 hour, bortezomib IV over 3 minutes, and dexamethasone IV or PO on days 1, 8, and 15. Patients also receive pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 8. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  cyclophosphamide: Given IV or PO
  pegylated liposomal doxorubicin hydrochloride: Given IV
  bortezomib: Given IV
  dexamethasone: Given IV or PO
Period: Overall Study
Arm/Group | Relapsed Disease (Cohort I) | Newly Diagnosed Disease (Cohort II)
Started | 6 | 25
Completed | 5 | 24
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor)
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of This Combination of Drugs as Assessed by the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (Cohort 1) [MTD Cyclophosphamide, MTD Bortezmib, MTD Docxorubicin]
Description: If 3 patients of cohort 1 require dose reduction of one or more of the medications for toxicity attributed to the drug or drugs, then the starting dose level will be reduced for that drug or drugs for future patients. The initial dosing of drugs for cohort 2 will be permitted to be one dose level above the maximal tolerated doses of cohort 1. Note that this Outcome Measure shows MTD for cyclophosphamide, bortezomib and doxorubicin. MTD for dexamethasone is include in a separate table due to the different Unit of Measure.
Time Frame: Up to 90 days after initiation of study treatment
Population: Patients with relapsed multiple myeloma who received cyclophosphomide, bortezomib, liposomal doxorubicin and dexamethasone. Note that the MTD for dexamethasone is in a separate table due to the different dosing unit.
Measure: Number; unit: mg/m2
Groups:
- Relapsed Disease: Patients with relapsed multiple myeloma receive cyclophosphamide IV or PO over 1 hour, bortezomib IV over 3 minutes, and dexamethasone IV or PO on days 1, 8, and 15. Patients also receive pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 8. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  cyclophosphamide: Given IV or PO
  pegylated liposomal doxorubicin hydrochloride: Given IV
  bortezomib: Given IV
  dexamethasone: Given IV or PO
Arm/Group | Relapsed Disease
Number analyzed (Participants) | 6
mg/m2
  MTD cyclophosphamide | 300
  MTD bortezomib | 1.6
  MTD liposomal doxorubicin | 30

2. Primary Outcome: Disease Response Rate (Cohort II)
Description: Disease response using Blade Multiple Myeloma Response Criteria in newly diagnosed (Cohort II) patients who completed at least one cycle of treatment. There were 24 evaluable patients in Cohort II.
Time Frame: up to 28 days after last cycle of treatment
Population: Newly diagnosed patients (cohort II)
Measure: Count of Participants; unit: Participants
Groups:
- Newly Diagnosed Patients: Patients with newly diagnosed multiple myeloma receive cyclophosphamide IV or PO over 1 hour, bortezomib IV over 3 minutes, and dexamethasone IV or PO on days 1, 8, and 15. Patients also receive pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 8. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  cyclophosphamide: Given IV or PO
  pegylated liposomal doxorubicin hydrochloride: Given IV
  bortezomib: Given IV
  dexamethasone: Given IV or PO
Arm/Group | Newly Diagnosed Patients
Number analyzed (Participants) | 24
Participants
  Complete response (CR) | 2
  Near complete response (nCR) | 2
  Very good partial response (VGPR) | 3
  Partial response (PR) | 11
  Stable disease (SD) | 6

3. Primary Outcome: Maximum Tolerated Dose of This Combination of Drugs as Assessed by the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (Cohort 1). [Dexamethasone MTD]
Description: If 3 patients of cohort 1 require dose reduction of one or more of the medications for toxicity attributed to the drug or drugs, then the starting dose level will be reduced for that drug or drugs for future patients. The initial dosing of drugs for cohort 2 will be permitted to be one dose level above the maximal tolerated doses of cohort 1. Note that this Outcome Measure will only describe the MTD for dexamethasone. Dexamethasone could not be reported with the MTD for the other three drugs due to a different Unit of Measure.
Time Frame: Up to 90 days after initiation of study treatment
Population: Patients with relapsed multiple myeloma who received cyclophosphomide, bortezomib, liposomal doxorubicin and dexamethasone. Note that this Outcome Measure will only describe the MTD for dexamethasone. Dexamethasone could not be reported with the MTD for the other three drugs due to a different Unit of Measure.
Measure: Number; unit: mg
Arm/Group | Relapsed Disease (Cohort I)
Number analyzed (Participants) | 6
mg | 40

ADVERSE EVENTS:
Time Frame: Through 45 days after the last dose of study drug.
Description: >= grade 2 events are recorded
Arm/Group | Treatment (Chemotherapy and Enzyme Inhibitor)
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy and Enzyme Inhibitor) (N=31)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy and Enzyme Inhibitor) (N=31)
Hand foot and mouth disease (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (2)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Acute exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Blistering hands (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Weight loss (Investigations) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 10 (10)
Constipation (Gastrointestinal disorders) | 10 (10)
Peeling hands (Skin and subcutaneous tissue disorders) | 1 (1)
Jaw pain (General disorders) | 1 (1)
Upper arm pain (General disorders) | 1 (1)
Fatigue (General disorders) | 18 (18)
Chest tightness (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Transaminitis (Investigations) | 1 (1)
Hypoalbuminemia (Investigations) | 5 (5)
Leg pain (General disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Vomiting (Eye disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 1 (1)
Skin changes (Skin and subcutaneous tissue disorders) | 1 (1)
Leukopenia (Investigations) | 4 (4)
Weakness (General disorders) | 1 (1)
Shoulder pain (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Back pain (General disorders) | 3 (3)
Neutropenia (Investigations) | 5 (5)
Hypophosphatemia (Investigations) | 3 (3)
Candidas (Infections and infestations) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Hypocalcemia (Investigations) | 3 (3)
Hiccoughs (General disorders) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphopenia (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days